CLINICAL TRIAL: NCT03629275
Title: A Randomized, Placebo-Controlled Study of the Efficacy and Safety of Intracerebral Stem Cells (CTX0E03) in Subjects With Disability Following an Ischemic Stroke
Brief Title: Investigation of Neural Stem Cells in Ischemic Stroke
Acronym: PISCES III
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic decision to progress stroke disability programme through regional partnerships
Sponsor: ReNeuron Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RN01-CP-0003
Record Dates: First submitted 2018-07-23; First posted 2018-08-14 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Ischemic Stroke; Chronic Stroke; Hemiparesis; Arm Paralysis
Keywords: Efficacy; Neural Stem cells; Intracerebral; Cerebral Infarction; Cerebrovascular disorders; Brain diseases; Stereotactic surgery
MeSH Terms: conditions — Ischemic Stroke; Paresis; Cerebral Infarction; Cerebrovascular Disorders; Brain Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- CTX0E03 Drug Product and delivery device (Experimental): 20 million neural stem cells
  Interventions: Combination Product: CTX0E03 Drug Product and delivery device
- Placebo (Sham Comparator): Sham Surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Combination Product: CTX0E03 Drug Product and delivery device — Includes stereotactic surgery and a burr hole drilled through the skull to allow for a one time intracerebral injection of 20 million CTX0E03 Drug Product stem cells into an area of the brain adjacent to the area affected by the stroke.
  Arms: CTX0E03 Drug Product and delivery device
Drug: Placebo — Sham surgical comparator includes stereotactic surgery and a partial thickness burr hole drilled into the skull. No injection of any kind is made into the brain, and no other intervention is given.
  Arms: Placebo

SUMMARY:
A study of stereotactic, intracerebral injection of CTX0E03 neural stem cells into patients with moderate to moderately severe disability as a result of an ischemic stroke.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, multi-center study. Patients with persistent disability 6-24 months following an ischemic stroke will be enrolled following confirmation of eligibility. Patients will be randomized 2:1 to undergo a stereotactic surgery and receive a single administration of CTX0E03 Drug Product by intracerebral implantation or undergo sham surgery only (placebo). Patients will be followed for 12 months after surgery with follow-up assessments occurring at various time points over the 12 months. All eligible patients will be assigned a standardized Physical Therapy (PT) program. Patients will complete their daily PT exercises at home for 12 weeks after their surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke that includes the supratentorial region as confirmed by CT or MRI, occurring within 6 to 24 months of the time that surgical intervention will be performed (Qualifying Stroke Event)
* Modified Rankin Score of 3 or 4 due to the Qualifying Stroke Event
* Some residual upper limb movement
* Sufficient cognitive and language abilities to comprehend verbal commands and to carry out the study assessments
* No medical conditions that would preclude neurosurgery with appropriate preparation and management.
* Ability to attend study visits and complete all study assessments including ability to provide informed consent

Exclusion Criteria:

* Modified Rankin Score of >1 prior to the Qualifying Stroke Event
* Stroke due to hemorrhage or stroke known or suspected of being caused by, or related to, connective tissue disorder, congenital disorder of the cerebral vessels or a disorder of thrombosis; patients with atrial fibrillation as a suspected cause of stroke are NOT excluded
* Neurosurgical pathway obstructed by vascular malformation or cavity
* History of neurological or other disease resulting in significant functional impairment (e.g. Parkinson's disease, motor neuron disease, moderate dementia, arthritis, contractures or fixed anatomical abnormality)
* Inability to stop or transition off valproic acid or other demethylating agents or Histone deacetylases (HDAC) inhibitors for 1 week before and 4 weeks after surgery
* Use of selective serotonin reuptake inhibitors (SSRI), unless the subject is on a stable dose that has been started at least 2-months before screening (V1)
* Use of antispasticity medications (excluding oral antispasticity medications if they have been taken regularly for at least one month prior to surgery)The use of Botox® or similar is allowed if the last dose was ≥3 months prior to screening; however, its use will be prohibited until following the 12 month visit
* Inability to discontinue anticoagulation therapy for a required interval
* History of malignant disease within the last 5 years, or any history of primary or secondary brain malignant disease
* Patients who have previously participated in a cell-based therapy study at any time or in any other study involving an investigational product or rehabilitation study within the last 30 days
* Patients with clinically significant lab values, including positive Class I human leukocyte antigen (HLA) antibodies specific for CTX0E03
* Planned initiation of any new PT regimen within 6-months of surgery

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects in which Modified Rankin Scale (mRS) improves by ≥1 point at Month 6 from Baseline | 6 months
  The mRS is an ordinal scale from 0-6, where 0 represents no disability, and each grade above 0 represents a subject's increased level of disability and dependence upon others to perform daily activities.

SECONDARY OUTCOMES:
Change from baseline in a subject's ability to execute activities of daily living using the Barthel Index (BI). | 6 months
  The BI is an ordinal scale used to measure a patient's ability to perform activities of daily living. Sum scores from 10 items are calculated with total possible scores ranging from 0-100, with lower scores indicating increased disability.
Change from baseline in a subject's basic mobility and balance using the Timed Up and Go Test (TUG). | 6 months
  TUG is a timed activity assessing mobility and balance in which subjects are asked to stand up from a chair, walk a distance of 3 meters, turn around, walk back to chair and seat themselves. Scores consist of time taken to complete the activity, in seconds.
Change from baseline in the function of subject's paretic limb using the Chedoke Arm and Hand Activity Inventory (CAHAI). | 6 months
  The CAHAI is validated to assess paretic limb function and consists of 13 functional tasks, each scored on a 7-point scale, with total test scores obtained by summing each task score. Total scores can range from 13-91 with higher scores indicating greater ability.
Change from baseline in a subject's executive processing speed, language skills and memory using the Symbol Digit Modalities Test. | 6 months
  Validated test assessing different aspects of cognitive function.
Change from baseline in a subject's executive processing speed, language skills and memory using Controlled Oral Word Association tasks. | 6 months
  Validated test assessing different aspects of cognitive function.
Change from baseline in a subject's executive processing speed, language skills and memory using the Multilingual Naming Test. | 6 months
  Validated test assessing different aspects of cognitive function.
Change from baseline in a subject's executive processing speed, language skills and memory using the Montreal Cognitive Assessment. | 6 months
  Validated test assessing different aspects of cognitive function.
Change from baseline in a subject's neurological deficits using the National Institute of Health Stroke Scale (NIHSS). | 6 months
  The NIHSS is comprised of 15 items used to assess severity of impairment due to stroke with each item scored on a 3 or 4 point ordinal scale in which 0 represents no impairment. Total sum score range from 0-42: higher score reflects greater severity.
Change from baseline in restoring a subject's motor function using the Fugl-Meyer Assessment of Motor Recovery after Stroke (FMA). | 6 months
  The FMA is used to assess motor function in post-stroke, hemiplegic patients. The FMA is comprised of 5 sections, and respective items within each section are scored using a 3-point ordinal scale with 0 representing inability to perform task. Total possible score is 226.
Change from baseline in subject's global rating of change regarding their limitations of activity, symptoms, and overall quality of life. | 6 months
  Self-administered 2 factor questionnaire assessing change in limitations of activity, symptoms, and overall quality of life.
Change from baseline in a subject's perception to stroke recovery using the Stroke Impact Scale (SIS). | 6 months
  The SIS is a stroke-specific, comprehensive measure of health status. The SIS is comprised of 59 items with each item rated on a 5 point Likert scale in terms difficulty. A score of 1 represents an inability to complete an item, where a score of 5 represents no difficulty.
Change from baseline in a subject's health-related quality of life using the EQ-5D-5L. | 6 months
  Subjects rate each of 5 dimensions with a numerical rating (1-5) where 1 represents no difficulty to 5 representing an inability, and where a lower total score represents better quality of life.
Safety: To assess the number and severity of adverse events and medical device incidents that occur over the study period. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Beckman, MD, Study Director — ReNeuron Ltd.
Locations (23):
- United States (23):
  - University of Arkansas, Little Rock, Arkansas
  - University of California, Irvine, Irvine, California
  - University of California, Los Angeles, Los Angeles, California
  - University of Southern California Neurorestoration Center, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California, San Diego, San Diego, California
  - University of Miami, Coral Gables, Florida
  - University of South Florida, Tampa, Florida
  - Emory, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Shirley Ryan Ability Lab, Chicago, Illinois
  - MedStar Health Research Institute, Hyattsville, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - JFK Neuroscience Institute, Edison, New Jersey
  - Albany Medical College, Albany, New York
  - Duke University School of Medicine, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Chattanooga Center for Neurologic Research, Chattanooga, Tennessee
  - University of Texas Health Science Center, Houston, Texas
  - University of Texas Health Science Center, San Antonio, Texas

REFERENCES:
- [Derived] Laskowitz DT, Muir KW, Savitz SI, Wechsler LR, Pilitsis JG, Rahimi SY, Beckman RL, Holmes V, Chen PR, Juel L, Koltai D, Kolls BJ. Methodological considerations in PISCES 3: a randomized, placebo-controlled study of intracerebral stem cells in subjects with disability following an ischemic stroke. Front Stroke. 2023 Jul 4;2:1182537. doi: 10.3389/fstro.2023.1182537. eCollection 2023. PMID 41541089
- [Derived] Kolls BJ, Muir KW, Savitz SI, Wechsler LR, Pilitsis JG, Rahimi S, Beckman RL, Holmes V, Chen PR, Albers DS, Laskowitz DT. Experience with a hybrid recruitment approach of patient-facing web portal screening and subsequent phone and medical record review for a neurosurgical intervention trial for chronic ischemic stroke disability (PISCES III). Trials. 2024 Feb 28;25(1):150. doi: 10.1186/s13063-024-07988-z. PMID 38419030
- [Derived] Olmsted ZT, Petersen EA, Pilitsis JG, Rahimi SY, Chen PR, Savitz SI, Laskowitz DT, Kolls BJ, Staudt MD. Toward Generalizable Trajectory Planning for Human Intracerebral Trials and Therapy. Stereotact Funct Neurosurg. 2022;100(4):214-223. doi: 10.1159/000521916. Epub 2022 Feb 7. PMID 35130557